CLINICAL TRIAL: NCT04900649
Title: Effect of Chest Resistance Exercise Combined With Chest Expansion Exercises on Respiratory Muscle Strength, Lung Function, and Thoracic Excursion in Children With Post-operative Congenital Diaphragmatic Hernia
Brief Title: Resistance Exercise in Children With Post-operative Congenital Diaphragmatic Hernia
Acronym: hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other); Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, College of Medical Rehabilitation, Qassim University, Saudi Arabia, Qassim, Buraidah. Consultant Physical Therapist, El-Sahel Teaching Hospital, General Organization for Teaching Hospitals and Institutes, Cairo, Egypt., Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/020/056
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Hernias, Diaphragmatic, Congenital
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): the study group has conducted chest resisted exercise combined with chest expansion exercise in addition to a usual chest physiotherapy. For chest resistance exercise, the children in the study group underwent sequential 12-week chest resistance exercise and chest expansion exercise, three sessions a week. Chest resistance exercises have been consisted of manual resistance exercise and resistance exercise via POWER breath KH2.
  Interventions: Other: chest resistance exercise
- control group (Experimental): 12-week usual chest physiotherapy in form of bilateral vibration and gentle percussion for 3-5 minutes with distal finger phalanges to the upper apical lobes in modified drainage positions, placing the patient in a side-lying position or a prone position to increase oxygenation, at least 2-3 times a week
  Interventions: Other: chest expansion exercises

INTERVENTIONS:
Other: chest resistance exercise — lung function.
  Other Names: respiratory muscle strength
  Arms: study group
Other: chest expansion exercises — thoracic excursion
  Other Names: POWER breath KH2
  Arms: control group

SUMMARY:
Congenital diaphragmatic hernia (CDH) is a life-threatening condition with long-term complications including respiratory tract infections, respiratory muscle weakness, and abnormal lung functions. This study, therefore, has been designed to ascertain the effect of chest resistance exercise and chest expansion exercise on respiratory muscle strength, lung function, and chest mobility in children with post-operative CDH.

DETAILED DESCRIPTION:
With the advances in surgical and neonatal treatment, the survival rates in children with CDH have been improved in the last decades. The surviving children may suffer from long-term complications such as impairments in lung growth (lung hypoplasia), cardiovascular disorders, pulmonary hypertension, gastrointestinal problems, and recurrent occurrence of lower respiratory tract infection. One of the physical therapy techniques used to treat chest disorders via encouraging the normal alignment of respiratory muscles with respiratory rhythm is chest resistance exercise through applying resistance to the sternal and coastal areas .

ELIGIBILITY:
Inclusion Criteria:

* ages between 10 and 14 years.
* the BMI between 20 and 25 Kg/m2. the children were considered as high risky CDH as they developed respiratory distress in the first days of their life.
* CDH was corrected surgically immediately after birth.
* children are still in following upstate in pediatric and physical therapy departments.

Exclusion Criteria:

* physical disability.
* diaphragmatic eventration.
* unable to perform all tests or procedures.
* children with cardiac anomalies

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle Strength | at baseline
  evaluated by using POWER breathe KH2 equipment.
Respiratory muscle Strength | after 12 weeks
  evaluated by using POWER breathe KH2 equipment.
Lung functions | at baseline
  assessed by the Minispir® Light spirometer with Winspiro® Light software. The child was seated with knees flexed 90° and was asked to hold three deep breaths, take deep inspiration to total lung capacity (TLC), then expire all the air inside the lungs to their residual volume (RV) to obtain the variables FEV1 (forced expiratory volume in 1 s) and FVC (forced vital capacity).
Lung functions | after 12 weeks
  assessed by the Minispir® Light spirometer with Winspiro® Light software. The child was seated with knees flexed 90° and was asked to hold three deep breaths, take deep inspiration to total lung capacity (TLC), then expire all the air inside the lungs to their residual volume (RV) to obtain the variables FEV1 (forced expiratory volume in 1 s) and FVC (forced vital capacity).

SECONDARY OUTCOMES:
Thoracic excursion | at baseline
  assessed by tape measurement
Thoracic excursion | after 12 weeks
  assessed by tape measurement

CONTACTS AND LOCATIONS:
Overall Officials: Walid Kamal, PhD, Study Chair — Prince Sattam Bin Abdulaziz University; Alshimaa Azab, PhD, Study Director — Cairo University
Locations (1):
- King Khalid Hospital, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Ackerman KG, Pober BR. Congenital diaphragmatic hernia and pulmonary hypoplasia: new insights from developmental biology and genetics. Am J Med Genet C Semin Med Genet. 2007 May 15;145C(2):105-8. doi: 10.1002/ajmg.c.30133. No abstract available. PMID 17436306
- [Result] Lally KP, Bagolan P, Hosie S, Lally PA, Stewart M, Cotten CM, Van Meurs KP, Alexander G; Congenital Diaphragmatic Hernia Study Group. Corticosteroids for fetuses with congenital diaphragmatic hernia: can we show benefit? J Pediatr Surg. 2006 Apr;41(4):668-74; discussion 668-74. doi: 10.1016/j.jpedsurg.2005.12.007. PMID 16567174
- [Result] Malaguti C, Rondelli RR, de Souza LM, Domingues M, Dal Corso S. Reliability of chest wall mobility and its correlation with pulmonary function in patients with chronic obstructive pulmonary disease. Respir Care. 2009 Dec;54(12):1703-11. PMID 19961637